CLINICAL TRIAL: NCT01497418
Title: Long Term Follow-up of the 23mm Portico™ Aortic Valve Implant and the SJM Transfemoral Delivery System
Brief Title: Long Term Follow-up of the 23mm Portico™ Aortic Valve Implant and the St. Jude Medical Transfemoral Delivery System
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 1102
Record Dates: First submitted 2011-12-02; First posted 2011-12-22 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Collect and evaluate the long term safety data.

DETAILED DESCRIPTION:
The purpose of this study is to collect and evaluate the long term safety data of the 23mm Portico™ Transcatheter Heart Valve and the transfemoral Delivery System previously implanted in subjects with aortic valve disease.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has given written study Informed Consent for participation prior to any study procedures.
2. Subject is ≥ 18 years of age or legal age in host country at time of consent.
3. Subject currently has a 23mm SJM Portico Transfemoral Transcatheter Heart Valve

Exclusion Criteria:

1. Subject currently participating in another investigational device or drug study.
2. Subject is unable or unwilling to return for the required follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that are candidate for implantation or have been implanted with the St. Jude Medical 23mm Portico Transcatheter heart valve.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2011-12; Primary Completion 2012-07 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The objective of this study is to retrospectively and prospectively collect and evaluate the long term safety of the 23mm Portico Transcatheter Aortic Heart | 1 year
  Data will be collected at 3 months, 6 months, and 12 months post-implant.

CONTACTS AND LOCATIONS:
Overall Officials: John Webb, MD, Principal Investigator — Providence Health Care - St. Paul's Hospital
Locations (2):
- Canada (2):
  - l'Institut universitaire de cardiologie et de pneumologie de Québec, Québec
  - St. Paul's Hospital, Vancouver